CLINICAL TRIAL: NCT06296784
Title: An E-health Psychoeducation Program to Manage Symptoms During COVID-19 Pandemic for People With Bipolar Disorders: a Randomized Controlled Study
Brief Title: An E-health Psychoeducation for People With Bipolar Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Collaborators: Alessandra Perra (Unknown)
Responsible Party: Principal Investigator, Mauro Giovanni Carta, Principal Investigator, University of Cagliari
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PG/2021/8551
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Bipolar Disorder; Psychoeducation; COVID-19 Pandemic
Keywords: Bipolar Disorder; Psychoeducation; COVID-19 Pandemic
MeSH Terms: conditions — Bipolar Disorder; COVID-19

STUDY DESIGN:
Intervention Model Description: Open-label cross-over randomized controlled trial (two arms)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-health psychoeducation (Experimental)
  Interventions: Other: e-health psychoeducation
- waiting list (No Intervention)

INTERVENTIONS:
Other: e-health psychoeducation — e-health psychoeducation intervention provides information about BD clinical condition and symptoms, as well as identifying effective coping strategies to manage symptoms and the dysregulation of biological rhythms. The content covered the impact of the pandemic and its related restrictions on mental health, particularly on anxiety and depressive symptoms. The intervention comprised one session per week for two months, and each session lasted approximately an hour and a half. It was conducted by healthcare professionals.
  Arms: e-health psychoeducation

SUMMARY:
This study aims to present data on the improvement of Quality of life (QoL), biological rhythms, anxiety, depressive symptoms and the correlations between QoL and biorhythms following an e-health psychoeducational intervention for Bipolar Disoirder (BD) during Covid-19 pandemic

DETAILED DESCRIPTION:
Biological rhythms significantly impact individuals' quality of life (QoL). During the COVID-19 pandemic, social rhythm dysregulation was identified as a contributing factor to relapses in Bipolar Disorder (BD). This trial aims to present data on the efficacy of an e-health psychoeducational intervention for BD in improving anxiety, depressive symptoms, QoL, biological rhythms, and the correlations between QoL and biorhythms.

This study employs a cross-over randomized controlled trial design. Inclusion criteria include a diagnosis of BD according to Diagnostic and Statistical Manual of mental disorders (DSM-V) criteria, age over 18, and obtaining informed consent.

The intervention consists of e-health psychoeducation aimed at reducing distress levels associated with the Covid-19 pandemic and the implemented restrictive measures (lockdown). The focus is on strategies to manage the dysregulation of biological rhythms, with one session per week over two months. Each session lasts approximately an hour and a half and is conducted by a team comprising psychologists, psychiatric rehabilitation technicians, and professional health educators.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of BD according to DSM-V, over 18 years old

Exclusion Criteria:

* do not have bipolar disorder, refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder (GAD-7) | T0 (0 weeks); T1 (8 weeks); T2 (16 weeks)
  GAD-7 is 7 item self-administered questionnaire evaluates symptoms of an anxiety disorder
Hamilton Depression Rating Scale (HDRS21) | T0 (0 weeks); T1 (8 weeks); T2 (16 weeks)
  Depressive symptoms were assessed using HDRS21 consists of 21 items, and the total score allows for the assignment of severity scores for the symptoms
Short Form Health Survey (SF-12) | T0 (0 weeks); T1 (8 weeks); T2 (16 weeks)
  SF12 is a self-administered questionnaire consisting of 12 items that assess two dimensions: physical health and mental health to establish poor/good QoL.
Biological Rhythms Interview of Assessment in Neuropsychiatry (BRIAN) | T0 (0 weeks); T1 (8 weeks); T2 (16 weeks)
  BRIAN is a interview consisting of 18 items that investigate four main areas related to the dysregulation of biological rhythms: sleeping, activity, social rhythms, and eating.

CONTACTS AND LOCATIONS:
Locations (1):
- San Giovanni di Dio Hospital, Cagliari, CA, Italy

IPD SHARING:
Plan to Share IPD: No